CLINICAL TRIAL: NCT01216618
Title: Evaluation of the Effect of the InsuPatch Device on Insulin Pharmacokinetics in Clamp Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G080106/A
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: MiniMed paradigm insulin pumps; insulin Lispro; Insulin Asprt.
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device (Experimental): Subject starts with two clamps including device use follows by a clamp without device use
  Interventions: Device: InsuPatch
- Control (No Intervention): Subject starts with clamps without device

INTERVENTIONS:
Device: InsuPatch — the InsuPatchTM device includes a heating pad and electronics. The heating pad is attached to an existing insulin infusion set by a simple procedure.
  Arms: Device

SUMMARY:
The study is a prospective, multi-center, open label, randomized; two-arms cross over study.

This is the test protocol for the InsuPatch device, whose purpose is to improve insulin delivery into the blood when the insulin is infused using an insulin-infusion pump by controlled heating of the area surrounding the point of infusion.

DETAILED DESCRIPTION:
Fifty five(55) type 1 IDDM subjects in three centers who use the MiniMed paradigm insulin pump, meeting the inclusion/exclusion criteria as outlined below and who provide written Informed Consent will be enrolled in the study.

The study will be done with subjects randomized into one of two procedure sequences. Each subject will undergo 3 procedures (two clamps with the InsuPatch and one clamp without the InsuPatch) and will thus serve as his/her own control. The same 55 subjects will be randomized into one sequence or the other. The order of the procedures will be selected randomly and will be performed both within one month.

There will be six Device visits starting with a screening and randomization visit, 3 clamps and a completion visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18- 65 years old (including = 18 years and =65 years)
2. Gender: men and women
3. BMI: 18-35 kg/m2
4. Type 1 Insulin dependent diabetes using the MiniMed paradigm insulin pumps for at least six months and using insulin Lispro or Insulin Aspart.
5. Diabetic subjects with HbA1c values below 9.5% (including 9.5%).
6. Subject understands the study requirements and the treatment procedures and has signed an Informed Consent before any study-specific tests or procedures are performed
7. Subject is willing to comply with all specified follow-up evaluations -

Exclusion Criteria:

1. Pregnancy
2. Breast feeding women.
3. Alcohol addiction
4. Had CABG (Coronary Artery Bypass Graft), are Post MI (Myocardial Infarction) or had active Ischemic heart disease prior to the study date
5. Had CVA (cardiovascular accident) or TIA (transient ischemic accident) prior to the study
6. Suffer from uncontrolled Hypertension (blood pressure in mm HG >160 systolic or > 95 diastolic)
7. Low blood hemoglobin concentration <9 g/dL for female and <11g/dL for male.
8. Abnormal kidney and/ or liver function tests. (If any of the liver or kidney function test parameters are greater than 3 fold normal values.
9. Subjects with Hyperthyroidism or Hypothyroidism with TSH level outside the normal range, TSH>5.5 mIU/L or TSH<0.4 mIU/L
10. Psychological incompetence
11. Any other clinical condition or history, that seems to be relevant to the principle investigator to disqualify the participant.
12. Subjects with diminished skin integrity
13. Subjects with heat sensitivity
14. Subjects involved in or planed to participate in other studies
15. Subjects using other drugs therapies to control blood glucose level other than insulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | Up to 5 hours
  Determination of insulin delivery to the blood as measured by Insulin levels in the blood derived from blood samples collected at pre-specified time points during the glucose clamp test.
Safety | Up to one month
  frequency and severity of all treatment-related adverse events until the completion of the study.

SECONDARY OUTCOMES:
pharmacokinetics | Up to 5 hours
  Cmax PK which is the highest concentration of insulin reached derived from blood samples collected at pre-specified time points during the glucose clamp test
Pharmacodynamic | Up to 5 hours
  Tmax PD which is the time of highest glucose infusion rate (GIR) derived from blood samples collected during the glucose clamp test

CONTACTS AND LOCATIONS:
Locations (3):
- Mills-Peninsula Health Services, San Mateo, California, United States
- Israel (2):
  - Wolfson Medical Center, Holon
  - Haddasah Medical Organization, Jerusalem

REFERENCES:
- See also: Sponsor's Official web site — http://www.insuline-medical.com